CLINICAL TRIAL: NCT00281489
Title: B-Unaware Study: Comparison of BIS-guided Anesthesia With End-Tidal Volatile-Guided Anesthesia to Decrease The Incidence of Awareness During High-Risk Surgery
Brief Title: Study Evaluating Ways of Preventing Patients From Being Awake During High-Risk Surgery and Anesthesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Michael Avidan, Director, Institute of Quality Improvement, Research & Informatics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-1112
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Explicit Recall of Intra-operative Events
Keywords: Recall; Awareness; BIS; Anesthesia; Explicit Recall

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- BIS Monitor guided algorithm (Experimental): BIS guided algorithm (BIS target 40 to 60) during anesthesia. Alarms when BIS is outside this range.
  Interventions: Device: BIS Monitor guided algorithm
- Volatile anesthetic guided algorithm (Active Comparator): Volatile anesthetic guided algorithm. Target anesthetic concentration 0.7 to 1.3 minimum alveolar concentration during anesthesia. Alarms when anesthetic concentration not in this range.
  Interventions: Behavioral: Volatile anesthetic guided algorithm

INTERVENTIONS:
Device: BIS Monitor guided algorithm — BIS guided algorithm (BIS target 40 to 60) during anesthesia. Alarms when BIS is outside this range.
  Arms: BIS Monitor guided algorithm
Behavioral: Volatile anesthetic guided algorithm — Volatile anesthetic guided algorithm. Target anesthetic concentration 0.7 to 1.3 minimum alveolar concentration during anesthesia. Alarms when anesthetic concentration not in this range.
  Arms: Volatile anesthetic guided algorithm

SUMMARY:
The overall purpose of this study is to see if a Bispectral Index (BIS) monitor, a Food and Drug Administration (FDA) approved brain monitoring device, will help to reduce the risk of patients remembering being awake during surgery. The BIS monitor may be able measure how asleep a patient is during surgery. Using the BIS monitor to guide anesthesia will be compared with using the concentration of anesthetic gas to guide anesthesia.

DETAILED DESCRIPTION:
General anesthesia is a state of drug-induced unconsciousness, during which patients should neither perceive nor recall noxious stimuli. Many patients facing surgery dread the prospect of being awake, in pain and unable to move owing to inadequate general anesthesia. A large multi-center study in the USA showed that, despite modern anesthesia techniques, the overall incidence of awareness or conscious recall remains about 0.1-0.2%. For high-risk (for awareness) surgery, such as cardiac surgery, trauma surgery and obstetric surgery, the incidence of conscious recall approaches 1%. This can lead to extreme anxiety and even posttraumatic stress disorder. Several monitors, including the Bispectral Index (BIS), which is based on processed electroencephalographic information, have been developed in an attempt to monitor depth of anesthesia. A recent landmark study suggested that harnessing the information provided by the BIS monitor decreases the incidence of explicit recall during high-risk surgical procedures from almost 1% to 0.1%. The possible impact of this study is enormous. The American Society of Anesthesiologists and the American Association of Nurse Anesthetists do not currently consider neurological monitors an essential part of routine anesthesia care. Increasingly, members of the anesthetic community are suggesting that for every patient undergoing general anesthesia, especially for procedures where the risk of awareness is considered higher, a neurological monitor, such as the BIS monitor, should be routinely applied.

Explicit recall under general anesthesia is a major concern among members of the public and has even been featured on the popular Oprah Winfrey Show. Several patients presenting for surgery at Barnes Jewish Hospital have questioned whether the anesthesia provider would be using a BIS monitor to "prevent awareness". Excluding the cost of the BIS monitor itself, the cost to use BIS is $17.50 for the disposable strip. If this monitor was to be used for every anesthetic administered at Barnes Jewish Hospital, this might translate to an annual cost of about $500,000. Explicit recall, especially when patients have been aware and unable to move, is a serious complication that frequently precipitates posttraumatic stress disorder. If indeed the BIS monitor does decrease the incidence of explicit recall, this could translate into a cost effective and more importantly clinically imperative intervention. Currently BIS monitors, or similar alternatives, are not used routinely to monitor depth of general anesthesia at Barnes Jewish Hospital.

However, there are several concerns regarding the studies that have been conducted using the BIS monitor. There have been no parameters guiding administration of anesthesia in the control groups. BIS data have not been collected for patients in control groups, which prevents retrospective analysis and assessment of the true sensitivity, specificity, positive and negative predictive values of the BIS recordings. Most of the studies have been funded by the manufacturer of the device, which introduces a potential conflict of interest and investigator bias. In view of the current pressure to adopt BIS monitoring or an equivalent into the standard of anesthesia care, it is essential to conduct a study to address some of the concerns. The hypothesis of this proposed study is that an anesthetic algorithm can be designed for high-risk surgical patients such that the incidence of awareness will be equivalent to or lower than that in a group where anesthesia depth is guided by the BIS monitor.

ELIGIBILITY:
Inclusion Criteria:

MUST HAVE:

General Anesthesia with volatile anesthetic

PATIENT CHARACTERISTICS

Major Criteria (any 1 of the following:)

1. Medications - anticonvulsants, abuse of opiates, benzodiazepines, cocaine
2. EF<40%
3. Prior history of awareness (recall)
4. History of difficult intubation or anticipated difficult intubation
5. ASA IV or V status
6. Aortic stenosis
7. End stage lung disease
8. Marginal exercise tolerance not secondary to musculoskeletal dysfunction
9. Pulmonary hypertension
10. Daily alcohol consumption

Minor Criteria (any 2 of the following)

1. Beta blockers
2. COPD
3. Moderate exercise tolerance not secondary to musculoskeletal dysfunction
4. Smokes ≥2 packs per day
5. Morbid obesity BMI>30 -

Exclusion Criteria:

1. Surgical procedure that prevents the use of the BIS (e.g surgery of forehead)
2. Patient positioning prevents use of the BIS
3. Surgery with wake-up test.
4. Less than 18 years of age
5. Vulnerable populations, such as those with dementia and those unable to provide informed consent.
6. Stroke with residual neurological deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The incidence of explicit recall of events during the surgical and anesthetic periods. | 30 days

SECONDARY OUTCOMES:
1 Anesthetic concentrations & BIS values in each group. | 1 day
2 Implicit memory (number). | 30 days
3 Dreaming. | 30 days
4 One-year mortality (and "anesthetic depth"). | 1 year
5 Relation of assessment to BIS value. | 30 days
6 Relation of events (e.g. movement) to BIS & ETAG. | 1 day
7 Relation of EMG to BIS. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine; Beth Burnside, Study Director — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Derived] Willingham M, Ben Abdallah A, Gradwohl S, Helsten D, Lin N, Villafranca A, Jacobsohn E, Avidan M, Kaiser H. Association between intraoperative electroencephalographic suppression and postoperative mortality. Br J Anaesth. 2014 Dec;113(6):1001-8. doi: 10.1093/bja/aeu105. Epub 2014 May 22. PMID 24852500
- [Derived] Avidan MS, Palanca BJ, Glick D, Jacobsohn E, Villafranca A, O'Connor M, Mashour GA; BAG-RECALL Study Group. Protocol for the BAG-RECALL clinical trial: a prospective, multi-center, randomized, controlled trial to determine whether a bispectral index-guided protocol is superior to an anesthesia gas-guided protocol in reducing intraoperative awareness with explicit recall in high risk surgical patients. BMC Anesthesiol. 2009 Nov 30;9:8. doi: 10.1186/1471-2253-9-8. PMID 19948045
- [Derived] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600